CLINICAL TRIAL: NCT05077917
Title: Cromolyn Sodium for Treatment of COVID-19 Pneumonia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Edward Michelson, MD, Professor and Chair, Dept of Emergency Medicine, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E21197
Record Dates: First submitted 2021-10-08; First posted 2021-10-14 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-05

CONDITIONS: COVID-19 Pneumonia; COVID-19 Respiratory Infection; Pneumonia, Viral
Keywords: COVID-19 pneumonia; Cromolyn sodium; Cromolyn
MeSH Terms: conditions — Pneumonia, Viral | interventions — Cromolyn Sodium; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled, randomized trial
Who Masked: Participant, Investigator
Masking Description: The participant, investigator, and the study team will be blinded to assignment of study drug or placebo. Only pharmacy and data committee will have key to drug assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cromolyn (Experimental): 2mL of 1% cromolyn sodium solution delivered via nebulizer 4 times a day for 4 days followed by 4% cromolyn solution administered intranasally 4 times per day for 14 days
  Interventions: Drug: Cromolyn Sodium
- Placebo (Placebo Comparator): 2-3mL of normal saline delivered via nebulizer 4 times a day for 4 days followed by intranasal administration of normal saline 4 times per day for 14 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cromolyn Sodium — Nebulized treatment for 4 days followed by intranasal treatment starting on day 5.
  Other Names: Nasal Crom
  Arms: Cromolyn
Other: Placebo — Nebulized treatment for 4 days followed by intranasal treatment starting on day 5.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The study hypothesis is that cromolyn, when combined with standard COVID-19 treatment, will improve patient symptoms and reduce the number of days to improved quality of life.

Investigators will study the effects of adding cromolyn to the standard treatment of hospitalized patients with COVID-19 pneumonia and who require supplemental oxygen. Cromolyn will be administered as a nebulized treatment four times a day for four days followed by intranasal administration for two weeks. Investigators may also screen for biomarkers that could indicate inflammatory responses and treatment-induced improvement.

Participants will receive either study drug or placebo which will be administered by nebulization for 4 days followed by 14 days of intranasal administration. Participants will be followed while in the hospital and then as outpatients up to day 21 following randomization.

DETAILED DESCRIPTION:
The study will take place in two phases: Phase 1 will be an open label study of 10 patients who will all receive the Cromolyn nebulization treatment followed by Cromolyn nasal spray to assess tolerability and response to the study treatment. Investigators may also draw blood from 10 healthy patients who will be the controls for the cellular and cytokine assays. Phase 2 will be a randomized double blind placebo-controlled study of 50 patients randomized 1:1 to receive Cromolyn nebulization followed by Cromolyn intranasal spray vs. saline nebulization and saline intranasal spray.

While subjects are hospitalized, investigators will record morning pulse, respiratory rate and oxygen saturation. Morning and daily peak oxygen supplementation as indicated by the use of high flow nasal cannula, non-invasive ventilation, or invasive ventilation will be recorded. The investigators will also note any improvement or decline in participant's condition and any reduction or increase in oxygen supplementation.

Follow-up phone calls (or EMR review if still hospitalized) will be made on days 7, 14, and 21 to assess dyspnea and physical function. Validated questionnaires from the Patient-Reported Outcomes Measurement Information System (PROMIS) (https://www.healthmeasures.net/explore-measurement-systems/promis) will be used to evaluate dyspnea and physical function. Once discharged, patients will also be asked to maintain a daily log of nasal drug use, COVID-19 symptoms, resting pulse and oxygen saturation which will be reviewed at the 21 day virtual visit.

ELIGIBILITY:
Inclusion Criteria:

1. COVID-19 symptoms (fever, cough, sore throat, malaise, headache, muscle pain, dyspnea at rest or with exertion, confusion, or respiratory distress),
2. diagnosis of COVID-19 pneumonia with an admission chest x-ray demonstrating multilobar ground glass infiltrates consistent with COVID-19 pneumonia.
3. room air estimated PaO2/FiO2 ratio between 150 -280
4. must correct to a pulse oximetry of 90% or better using no more than 5 liters of low flow supplemental oxygen
5. must be enrolled within 24 hours of hospital admission

Exclusion Criteria:

1. immunocompromised due to current use of immunosuppressive drugs or chemotherapy, have a history of HIV/organ transplant/ active hepatitis B or C, or are on hemodialysis or peritoneal dialysis
2. currently on oxygen supplementation greater than low flow nasal cannula (including home oxygen therapy; CPAP for obstructive sleep apnea is not an exclusion)
3. have DNR status or not expected to survive >7 days
4. experiencing shock (on vasopressors) or multiple organ dysfunction or failure
5. are co-infected with influenza A or B
6. history of DVT or PE within last 12 weeks
7. currently pregnant or nursing
8. participating in another therapeutic trial
9. allergic to cromolyn sodium.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Change in requirement for oxygen supplementation based on daily assessment of flow (LPM or %Fi O2) and delivery device (cannula, mask, CPAP/BiPAP, ventilator) | up to 21 days
  Determination of trend in subject's need for oxygen supplementation over time.
Change in respiratory symptoms (cough, shortness of breath, and fatigue) determined by data extraction from medical record, self-assessment by subject, or subject survey as appropriate for stage of the study. | up to 21 days
  Determination of trend in subject's respiratory symptoms over time.

SECONDARY OUTCOMES:
hospital length of stay | up to 21 days
  number of days from admission to discharge
change the patient score from the PROMIS survey provided to subjects at days 7, 14, and 21. | up to 21 days
  Determination of number of days to improved quality of life (QOL) from start of study treatment

OTHER OUTCOMES:
number of return visits to hospital | up to 21 days
  any readmission to hospital after discharge
assignment of COVID-19 outcomes | up to 21 days
  based on WHO classification

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Michelson, MD, Principal Investigator — Texas Tech University Health Sciences Center, Department of Emergency Medicine
Locations (1):
- University Medical Center of El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No